CLINICAL TRIAL: NCT04542928
Title: Effectiveness of a Nurse Facilitated Face Care Group in Patients With Schizophrenia：A Randomized Controlled Trial
Brief Title: Effectiveness of a Nurse Facilitated Face Care Group in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSPH-2019-17
Record Dates: First submitted 2020-04-19; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-07

CONDITIONS: Body Image

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine care (Placebo Comparator): The controlled group will receive routine functional treatment activities, a facial cleansing instruction and five facial cleansing videos.
  Interventions: Behavioral: nurse facilitated face care group
- experimental group (Experimental): experimental group is required to receive a nurse leading 50- minute face care group every two weeks
  Interventions: Behavioral: nurse facilitated face care group

INTERVENTIONS:
Behavioral: nurse facilitated face care group — The experimental group is required to receive a nurse leading 50- minute face care group every two week

SUMMARY:
This study aims to explore the effectiveness of nurse-facilitated face care group on body image and self-esteem in female patients with schizophrenia.

DETAILED DESCRIPTION:
Many studies have shown that patients with schizophrenia have poor cleanliness and negligible appearance, which leads to negative body image and low self-esteem. However, there are few researches in Taiwan that nurse facilitated face care group in patients with schizophrenia to improve their body image and self-esteem.This study was to explore the effectiveness of a nurse facilitated face care group in patients with schizophrenia in improving their body image and self-esteem.A total of 96 patients with schizophrenia in a mental hospital in southern Taiwan were recruited in this study. The participants were divided into experimental and control groups through block randomization. In addition to participating in routine functional treatment activities, the experimental group is required to receive an additional 50 minutes of face care grou every two weeks led by the nurse. The patients in control group received routine functional treatment activities, a facial cleansing instruction and five facial cleansing videos. The research tools include demographic data, the subscale in MBSRQ - Appearance evaluation and Appearance orientation, FACE-Q - Appearance-related psychosocial distress. FACE-Q - Satisfaction with outcome. FACE-Q - Psychological function. FACE-Q - Satisfaction with skin. FACE-Q - Social function. Rosenberg self-Esteem scale (RSES). A questionnaire survey of body image and self-esteem was conducted before the intervention, 12 weeks after the intervention and one month after the end of the intervention.The collected data were analyzed by IBM SPSS 24.0 statistical software. The descriptive statistics include mean, minimum, maximum, standard deviation, frequency distribution, and percentages; the Generalized estimating equation (GEE) were employed to explore the effectiveness of a nurse facilitated face care group in patients with schizophrenia after controlling demographic data.

ELIGIBILITY:
Inclusion Criteria:

* People with Schizophrenia and schizoaffective disorder for more than two years.
* The age is above 20 year.
* Can communicate with Mandarin or Taiwanese.
* The score of the Positive and Negative Syndrome Scale(PANSS) is below 60(included).
* People are willing to participate in this study, can read and know the consent and can sign on the consent by their own.

Exclusion Criteria:

* Exclude people with a personality disorder, brain injury, cognitive impairment, Intellectual Developmental Disorder or substance use disorder.
* people who are not willing to sign the consent.
* people can not read.
* people can not communicate with Mandarin or Taiwanese.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 97 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-07-12 (Actual); Study Completion 2020-07-25 (Actual)

PRIMARY OUTCOMES:
Change in FACE-Q - Appearance-related psychosocial distress | pre-intervention(T0), at 12 weeks (T1) and 16 weeks (T2)
  To measure the level of Appearance-related psychosocial distress.There are 8 items in this scale. Using Likert scale to rate each item (1=Strongly disagree, 2=disagree, 3=agree, 4=strongly agree).Higher scores reflect more appearance-related psychosocial distress.
Change in FACE-Q - Satisfaction with outcome | pre-intervention(T0), at 12 weeks (T1) and 16 weeks (T2)
  To measure satisfaction with outcome.There are 6 items in this scale. Using Likert scale to rate each item (1=Strongly disagree, 2=disagree, 3=agree, 4=strongly agree).Higher scores reflect more satisfaction with outcome.
Change in The Appearance evaluation subscale in MBSRQ | pre-intervention(T0), at 12 weeks (T1) and 16 weeks (T2)
  To measure the attractiveness or lack of attractiveness of an individual's physical appearance, a person's satisfaction or dissatisfaction with his appearance.There are 7 items in this scale. Using Likert scale to rate each item (1=Strongly disagree, 2=disagree, 3=neither agree nor disagreeagree, 4=agree, 5=strongly agree).Higher scores reflect more satisfied you are with your appearance
Change in The Appearance orientation subscale in MBSRQ | pre-intervention(T0), at 12 weeks (T1) and 16 weeks (T2)
  To assess how much the individual attaches importance to appearance.There are 12 items in this scale. Using Likert scale to rate each item (1=Strongly disagree, 2=disagree, 3=neither agree nor disagreeagree, 4=agree, 5=strongly agree).Higher scores reflect more you care about your appearance.
Change in FACE-Q -Psychological function | pre-intervention(T0), at 12 weeks (T1) and 16 weeks (T2)
  To measure psychological function.There are 10 items in this scale. Using Likert scale to rate each item (1=Strongly disagree, 2=disagree, 3=agree, 4=strongly agree).Higher scores reflect higher psychological function.
Change in FACE-Q -Satisfaction with skin | pre-intervention(T0), at 12 weeks (T1) and 16 weeks (T2)
  To measure satisfaction with skin.There are 12 items in this scale. Using Likert scale to rate each item (1=Strongly disagree, 2=disagree, 3=agree, 4=strongly agree).Higher scores reflect more satisfaction with skin.
Change in FACE-Q -Social function | pre-intervention(T0), at 12 weeks (T1) and 16 weeks (T2)
  To measure satisfaction with skin.There are 8 items in this scale. Using Likert scale to rate each item (1=Strongly disagree, 2=disagree, 3=agree, 4=strongly agree).Higher scores reflect higher social function.

SECONDARY OUTCOMES:
Change in Rosenberg self-Esteem scale (RSES) | pre-intervention(T0), at 12 weeks (T1) and 16 weeks (T2)
  To measure the level of self-esteem.There are 10 items in this scale. Using Likert scale to rate each item (1=Strongly disagree, 2=disagree, 3=agree, 4=strongly agree) and higher score means higher level of self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Tu-Lin Lin, BSN, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan